CLINICAL TRIAL: NCT03436420
Title: Gemcabene for the Treatment of Pediatric NAFLD: A Phase 2a Study
Brief Title: Gemcabene for the Treatment of Pediatric NAFLD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to lack of efficacy and safety concerns.
Sponsor: Emory University (Other)
Collaborators: Gemphire Therapeutics (Industry)
Responsible Party: Principal Investigator, Miriam Vos, MD, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00099844
Record Dates: First submitted 2018-02-11; First posted 2018-02-19 (Actual); Results first posted 2020-11-12 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Pediatrics; Lipids; Liver Diseases; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Obesity | interventions — gemcabene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gemcabene (Experimental): Children receiving 12 weeks of treatment with gemcabene
  Interventions: Drug: Gemcabene

INTERVENTIONS:
Drug: Gemcabene — Participants will take 300 milligrams (mg) of gemcabene, once per day for 12 weeks.
  Other Names: Gemcabene calcium

SUMMARY:
This is a multicenter, prospective, open-label, Phase 2, proof of concept study to test preliminary efficacy and safety of gemcabene in children with established nonalcoholic fatty liver disease (NAFLD) incompletely treated by lifestyle changes. The hypothesis of the study is that 300 mg of gemcabene once a day for 12 weeks will reduce alanine aminotransferase (ALT), hepatic steatosis, dyslipidemia and down regulate de novo lipogenesis in children with NAFLD.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) has quickly become the most common liver disease in children in the US and is rising worldwide. While the true prevalence and incidence are not known, estimates have placed prevalence in the US as high as 7 million children. The prevalence varies greatly across race and ethnic groups with Hispanic, Asian and White children having increased rates compared to African American children. Lifestyle changes are the first line treatment, but many children fail to respond to these. Pharmaceutical treatments are needed for children that cure NAFLD and ideally also benefit the systemic features (dyslipidemia, insulin sensitivity, BMI). Gemcabene calcium (Gemcabene) is a promising therapeutic that may benefit pediatric NAFLD and early phase trials are needed to support further development for this indication. It has several mechanisms of action including enhancing the clearance of very-low-density lipoprotein (VLDL) and blocking the production of hepatic triglyceride and cholesterol synthesis. Gemcabene was previously tested in adults for treatment of dyslipidemia and has extensive safety data.

In this study, 40 children ages 12-17 years with histologically confirmed NAFLD or MRI based diagnosis and elevated ALT will receive 300 mg of gemcabene per day for 12 weeks. Study visits will occur at screening, baseline, week 2, week 6 and week 12. A follow up phone call will occur one month after the child stops taking the study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Provision of signed and dated assent, if indicated
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. Children aged 12-17 years at the time of informed consent
5. History of clinical diagnosis of NAFLD including a, b and c below:

   1. Medical history eliminating, other chronic liver diseases (for example mitochondrial diseases, hepatotoxic drugs, anorexia nervosa)
   2. Laboratory studies: negative testing for hepatitis C and normal ceruloplasmin
   3. Either liver biopsy confirming NAFLD or MRI > 10% steatosis within the past three years
6. ALT ≥ 54 U/L for boys or ≥ 46 U/L for girls and ≤ 250 U/L at screening visit and within past three months (prior to screening). If ALT at screening is more than two times the historic value (or a historic value is not available), the subject will be asked to repeat the ALT after four weeks. If the repeat ALT is more than 50% increased or decreased over the screening ALT a third ALT may be obtained. If a third ALT is not within 50% of the previous value then the subject is ineligible, but may be rescreened at a later date.
7. Body weight ≥ 60 kg at the time of screening
8. Able to take oral medication and be willing to adhere to the study drug regimen
9. Minimum of three months of attempted lifestyle modification to treat the NAFLD and agreement to adhere to Lifestyle Considerations (dietary improvement and physical activity) throughout study duration

Exclusion Criteria:

1. Heart disease (e.g., myocardial infarction, heart failure, unstable arrhythmias)
2. Seizure disorder
3. Active coagulopathy (international normalized ratio (INR) > 1.4)
4. Renal dysfunction with an estimated glomerular filtration rate (eGFR) <60ml/min/1.73 calculated using Schwartz Bedside GFR calculator for children
5. History of active malignant disease requiring chemotherapy or radiation
6. History of significant alcohol intake (AUDIT questionnaire) or inability to quantify alcohol consumption
7. Use of new medications or supplements with the intent to treat NAFLD/nonalcoholic steatohepatitis (NASH) during the 30 days prior to screening, including statin therapy. Medications or supplements (including metformin and vitamin E) that they have been on and are on a stable dose are acceptable
8. History of bariatric surgery or planning to undergo bariatric surgery during study duration
9. Clinically significant depression
10. Any girl nursing, planning a pregnancy, known or suspected to be pregnant, or who has a positive pregnancy screen
11. Non-compensated liver disease defined as cirrhosis and any one of the following hematologic, biochemical, and serological criteria on entry into protocol:

    * Hemoglobin < 10 g/dL;
    * White blood cell (WBC) < 3,500 cells/mm3;
    * Neutrophil count < 1,500 cells/mm3;
    * Platelets < 150,000 cells/mm3;
    * Total bilirubin > 1.3 mg/dL unless due to Gilbert's syndrome (subjects with a history of Gilbert's syndrome may be included if both direct bilirubin and the reticulocyte count do no exceed the upper limit of normal (ULN) [reflexive direct bilirubin testing will be used to confirm Gilbert's syndrome])
    * Albumin < 3.2 g/dL
    * INR > 1.3
    * Abnormal alkaline phosphatase
    * Any history of ascites, variceal bleeding, hepatic encephalopathy, or hepatocellular carcinoma (HCC)
12. Poorly controlled diabetes mellitus (hemoglobin A1c (HbA1c) > 8%) or requiring insulin
13. Patients with type I diabetes mellitus
14. Chronic liver disease other than NAFLD
15. Patients on Cytochrome P450 3A4 (CYP3A4) inhibitors such as itraconazole or macrolide antibiotics are excluded
16. Patients who are on thiazolidinediones, fibrates or fish oils are excluded
17. Patients who are on daily prescription medications are excluded except for allergy medications, Attention Deficit Hyperactivity Disorder (ADHD) medications, asthma medications, or any other acceptable medication in the opinion of the investigator
18. Abnormal creatinine kinase levels at screening (may be repeated if the elevation is thought to be exercise related)
19. Sexually active female participants of childbearing potential and Tanner stage ≥ 4 or menstruating unwilling to utilize two acceptable forms of contraception from screening through completion of the study or unwilling to complete pregnancy tests throughout the study
20. Currently enrolled in a clinical trial or who received an investigational study drug within 90 days of screening
21. Participants who are not able or willing to comply with the protocol or have any other condition that would impede compliance or hinder completion of the study, in the opinion of the investigator

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam B Vos, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta / Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were recruited from the patient population of Children's Healthcare of Atlanta, in Atlanta, Georgia. Enrollment began on March 29, 2018 and study follow up was completed on August 27, 2019.
Groups:
- Gemcabene: Children with nonalcoholic fatty liver disease (NAFLD) receiving 12 weeks of treatment with gemcabene
Period: Overall Study
Arm/Group | Gemcabene
Started | 6
Completed | 3
Not Completed | 3
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Population: The baseline analysis includes all children who began the trial.
Groups:
- Gemcabene: Children with NAFLD receiving 12 weeks of treatment with gemcabene
Arm/Group | Gemcabene
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Alanine Aminotransferase (ALT)
Description: Percent change in alanine aminotransferase (ALT) from baseline to 12 weeks was examined. ALT elevation is the most common screening test used for detecting NAFLD. The normal range for ALT varies by age, sex, and the specific assay used but is approximately 9-23 units/Liter (U/L) for boys and girls aged 1-18. Children with a sustained ALT ≥ 80 U/L are twice as likely to have nonalcoholic steatohepatitis (NASH), which is a severe form of NAFLD characterized by inflammation and liver cell damage.
Time Frame: Baseline, Week 12
Population: This analysis includes participants completing 12 weeks of gemcabene.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
Percent change | 79.86 (27.02)

2. Secondary Outcome: Absolute Change in ALT
Description: Absolute change in ALT among study participants is reported here. ALT elevation is the most common screening test used for detecting NAFLD. ALT elevation is the most common screening test used for detecting NAFLD. The normal range for ALT varies by age, sex, and the specific assay used but is approximately 9-23 U/L for boys and girls aged 1-18. Children with a sustained ALT ≥ 80 U/L are twice as likely to have nonalcoholic steatohepatitis (NASH), which is a severe form of NAFLD characterized by inflammation and liver cell damage.
Time Frame: Baseline, Week 6, Week 12
Population: This analysis includes participants who completed the trial up to Week 6 or Week 12.
Measure: Mean (Standard Deviation); unit: Units/Liter (U/L)
Arm/Group | Gemcabene
Number analyzed (Participants) | 4
Units/Liter (U/L)
  Baseline to Week 6 | 55.50 (49.55)
  Baseline to Week 12: number analyzed (Participants) | 3
  Baseline to Week 12 | 80.33 (63.26)

3. Secondary Outcome: Percent Change in ALT Between Study Visits
Description: Percent change in ALT from baseline to week 6 and the mean of week 6 and week 12 was examined. ALT elevation is the most common screening test used for detecting NAFLD. The normal range for ALT varies by age, sex, and the specific assay used but is approximately 9-23 U/L for boys and girls aged 1-18. Children with a sustained ALT ≥ 80 U/L are twice as likely to have nonalcoholic steatohepatitis (NASH), which is a severe form of NAFLD characterized by inflammation and liver cell damage.
Time Frame: Baseline, Week 6, Week 12
Population: This analysis includes participants who completed the trial up to Week 6 or Week 12.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Gemcabene
Number analyzed (Participants) | 4
Percent change
  Baseline to Week 6 | 58.47 (48.90)
  Week 6 to Week 12: number analyzed (Participants) | 3
  Week 6 to Week 12 | 4.58 (12.31)

4. Secondary Outcome: Absolute Change in Hepatic Steatosis
Description: Hepatic steatosis (fat accumulation in the liver) was measured by MRI using liver fat fraction (HepaFat-Scan by Resonance Health). NAFLD is characterized by an accumulation of fat in the liver. Having a fat percentage greater than 5% of the weight of the liver is a typical cut point to indicate NAFLD. The HepaFat-Scan software is a non-invasive method of measuring the volumetric liver fat fraction and is validated in children.
Time Frame: Baseline, Week 12
Population: This analysis includes participants completing 12 weeks of gemcabene.
Measure: Mean (Standard Deviation); unit: percentage of fat
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
percentage of fat | 9.87 (4.06)

5. Secondary Outcome: Absolute Change in Pancreatic Fat
Description: Pancreatic fat was measured by MRI (HepaFat). Increased pancreatic fat is associated with more severe liver disease in children with NAFLD.
Time Frame: Baseline, Week 12
Population: This analysis includes participants completing 12 weeks of treatment.
Measure: Mean (Standard Deviation); unit: percentage of fat
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
percentage of fat | 2.70 (2.26)

6. Secondary Outcome: Absolute Change in Aspartate Aminotransferase (AST)
Description: AST is a common screening test used for detecting NAFLD. The normal range for AST varies by age, sex, and the specific assay used but is approximately 13-32 U/L for boys and 12-24 units/Liter for girls aged 7-18. Elevated AST levels indicate increased liver disease.
Time Frame: Baseline, Week 6, Week 12
Population: This analysis includes participants who completed the trial up to Week 6 or Week 12.
Measure: Mean (Standard Deviation); unit: Units/Liter (U/L)
Arm/Group | Gemcabene
Number analyzed (Participants) | 4
Units/Liter (U/L)
  Baseline to Week 6 | 17.25 (12.15)
  Baseline to Week 12: number analyzed (Participants) | 3
  Baseline to Week 12 | 30.33 (23.38)

7. Secondary Outcome: Change in Fasting Insulin
Description: Insulin sensitivity was determined by assessment of fasting insulin. Fasting insulin increases with insulin resistance and tends to occur with NAFLD.
Time Frame: Baseline, Week 6, Week 12
Population: This analysis includes participants who completed the trial up to Week 6 or Week 12 and who had their blood sample analyzed.
Measure: Mean (Standard Deviation); unit: micro international unit per mL (uIU/mL)
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
micro international unit per mL (uIU/mL)
  Baseline to Week 6 | 5.73 (16.22)
  Baseline to Week 12 | 16.03 (20.93)

8. Secondary Outcome: Change in Fasting Glucose
Description: Insulin sensitivity was determined by assessment of fasting glucose. The normal range for fasting glucose in children is 70-99 mg/dL. Diabetes mellitus is indicated with fasting glucose levels of 126 or greater.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
milligrams per deciliter (mg/dL)
  Baseline to Week 6 | -1.03 (9.65)
  Baseline to Week 12 | -2.63 (1.40)

9. Secondary Outcome: Change in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) Score
Description: The HOMA-IR score is calculated as fasting blood glucose level (nmol/L) multiplied by fasting insulin level (microU/L), divided by 22.5. Higher scores indicate increasing insulin resistance, although pediatric cut-points for HOMA-IR scores vary by gender and age.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
units on a scale
  Baseline to Week 6 | 1.11 (4.32)
  Baseline to Week 12 | 3.75 (5.38)

10. Secondary Outcome: Absolute Change in Gamma-glutamyltransferase (GGT)
Description: Gamma-glutamyl transferase (GGT) is a biomarker for NAFLD. Normal GGT values vary by age and the specific assay used. The normal range for males and females aged 11-18 is approximately 5-15 U/L. Increased GGT is associated with more severe NAFLD.
Time Frame: Baseline, Week 6, Week 12
Population: This analysis includes participants who completed the trial up to Week 6 or Week 12.
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Gemcabene
Number analyzed (Participants) | 4
International units per liter (IU/L)
  Baseline to Week 6 | 2.00 (3.16)
  Baseline to Week 12: number analyzed (Participants) | 3
  Baseline to Week 12 | 6.67 (2.31)

11. Secondary Outcome: Absolute Change in Total Cholesterol
Description: Blood was drawn for a clinical lipid profile, including total cholesterol. Cholesterol is waxy substance which is produced by the liver or comes from food consumed. Cholesterol concentrations are commonly used as a marker for cardiovascular disease risk in adulthood Total cholesterol levels below 170 mg/100 milliliters (mL) of blood are in the normal range while levels at 200 and above are considered high.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
mg/dL
  Baseline to Week 6 | -4.00 (17.78)
  Baseline to Week 12 | -2.33 (15.31)

12. Secondary Outcome: Absolute Change in Non-high-density Lipoprotein Cholesterol (Non-HDL-C)
Description: Blood was drawn for a clinical lipid profile, including total non-HDL-C. A measurement of non-HDL-C is obtained by subtracting high-density lipoprotein (HDL) level from total cholesterol. Non-HDL-C can predict atherosclerosis with as much accuracy as other lipoproteins can. Non-HDL-C values of 129 mg/dL or greater are considered high.
Time Frame: Baseline, Week 6, Week 12
Population: This analysis was not performed due to early termination of the study. Frozen samples were to be run in batches upon completion of the study, however, very few samples had been collected as the study did not reach completion. As the milestones for study completion were not met, funding for running the samples was not available.
Arm/Group | Gemcabene
Number analyzed (Participants) | 0

13. Secondary Outcome: Absolute Change in High-density Lipoprotein (HDL) Cholesterol
Description: Blood was drawn for a clinical lipid profile, including total HDL cholesterol. HDL cholesterol is the "good" cholesterol because it is a type of fat that removes cholesterol from blood, thereby preventing build up. A healthy value for HDL cholesterol is 35 mg/dL and higher. Values under 35 mg/dL mean the child has a higher risk of developing heart disease.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
milligrams per deciliter (mg/dL)
  Baseline to Week 6 | -1.97 (2.55)
  Baseline to Week 12 | -2.97 (4.96)

14. Secondary Outcome: Absolute Change in Very-low-density Lipoprotein Cholesterol (VLDL-C)
Description: Blood was drawn for a clinical lipid profile, including total VLDL cholesterol. VLDL cholesterol is produced in the liver and high levels are associated with increased plaque buildup in arteries. Values of VLDL-C that are 29 mg/dL or greater are considered high.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 12
Arm/Group | Gemcabene
Number analyzed (Participants) | 0

15. Secondary Outcome: Absolute Change in Low-density Lipoprotein (LDL) Cholesterol
Description: Blood was drawn for a clinical lipid profile, including LDL cholesterol. LDL cholesterol levels below 110 mg/100 mL of blood are in the normal range while levels at 130 and above are considered high.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
milligrams per deciliter (mg/dL)
  Baseline to Week 6 | -1.33 (18.88)
  Baseline to Week 12 | -2.67 (12.74)

16. Secondary Outcome: Absolute Change in Triglycerides (TG)
Description: Blood was drawn for a clinical lipid profile, including triglycerides. Triglycerides are made by the body and come from food consumed. High triglyceride levels increases the risk of heart disease and stroke. Triglyceride levels below 150 mg/dL are considered acceptable while levels greater than 200 mg/dL are considered high.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
milligrams per deciliter (mg/dL)
  Baseline to Week 6 | -7.33 (41.31)
  Baseline to Week 12 | 31.67 (7.64)

17. Secondary Outcome: Absolute Change in Apolipoprotein A-1 (ApoA-1)
Description: Apolipoproteins transport lipids through the body by binding with fat and cholesterol to form lipoproteins. ApoA-1 is a component of HDL ("good cholesterol") which transports cholesterol and phospholipids through the body to the liver. Among children aged 2 to 17 years, an ApoA-1 level of less than 115 mg/dL is considered low and levels greater than 120 mg/dL are considered acceptable.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
milligrams per deciliter (mg/dL)
  Baseline to Week 6 | -2.27 (10.27)
  Baseline to Week 12 | 0.80 (15.09)

18. Secondary Outcome: Absolute Change in Apolipoprotein B (ApoB)
Description: Apolipoproteins transport lipids through the body by binding with fat and cholesterol to form lipoproteins. ApoB is a component of VLDL, intermediate-density lipoproteins (IDL), LDL, and chylomicrons. Among children aged 2 to 17 years, an ApoB level of less than 90 mg/dL is considered acceptable and levels of 100 mg/dL and greater are considered high.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
milligrams per deciliter (mg/dL)
  Baseline to Week 6 | 0.90 (15.02)
  Baseline to Week 12 | 3.07 (8.19)

19. Secondary Outcome: Absolute Change in Apolipoprotein C-II (ApoC-II)
Description: Apolipoproteins transport lipids through the body by binding with fat and cholesterol to form lipoproteins. ApoC-II is a component of VLDL and chylomicrons. Normal values are between 3-5 mg/dL and abnormal values may be caused by a lipoprotein lipase deficiency resulting in fats not being broken down normally. Abnormal ApoC-II measurements may explain elevated levels of cholesterol and triglycerides.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
milligrams per deciliter (mg/dL)
  Baseline to Week 6 | 0.03 (0.89)
  Baseline to Week 12 | 0.95 (0.58)

20. Secondary Outcome: Absolute Change in Apolipoprotein E (ApoE)
Description: Apolipoproteins transport lipids through the body by binding with fat and cholesterol to form lipoproteins. ApoE is a component of IDL and chylomicrons and carry cholesterol to the brain. Normal values of ApoE are between 3-7 mg/dL. Elevated ApoE may be associated with increased risk of dyslipidemia and atherosclerosis.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
milligrams per deciliter (mg/dL)
  Baseline to Week 6 | 0.24 (0.54)
  Baseline to Week 12 | 0.26 (0.11)

21. Secondary Outcome: Absolute Change in Apolipoprotein CIII (ApoCIII)
Description: Apolipoproteins transport lipids through the body by binding with fat and cholesterol to form lipoproteins. ApoCIII is a component of VLDL, HDL, and triglyceride-rich chylomicrons and regulates lipid metabolism. Elevated ApoCIII is associated with atherosclerosis and cardiovascular disease.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
mg/dL
  Baseline to Week 6 | -1.80 (2.59)
  Baseline to Week 12 | 0.87 (0.96)

22. Secondary Outcome: Absolute Change in High Sensitivity C-Reactive Protein (hsCRP)
Description: High Sensitivity C-Reactive Protein (hsCRP) is a measurement assessing inflammation. Increased levels of hsCRP are associated with increased risk of cardiovascular disease or cardiovascular events such as stroke or heart attack. Values of hsCRP that are less than 1.0 mg/L are considered low risk, 1.0 to 3.0 mg/L indicates average risk, and values greater than 3.0 mg/L are considered high risk.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
milligrams per liter (mg/L)
  Baseline to Week 6 | 0.21 (0.15)
  Baseline to Week 12 | 1.15 (1.42)

23. Secondary Outcome: Change in Interleukin 1 Beta (IL-1B)
Description: Interleukin 1 beta is a cytokine protein involved in inflammatory response. A normal value for IL-1B is less than 3.9 picograms per milliliter (pg/mL). Increased IL-1B levels have been found to be associated with congestive heart failure.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 12
Arm/Group | Gemcabene
Number analyzed (Participants) | 0

24. Secondary Outcome: Change in Interleukin 6 (IL-6)
Description: Interleukin 6 is a cytokine protein involved in the pro-inflammatory and anti-inflammatory response and stimulates an inflammatory response in many diseases, including atherosclerosis. Higher levels are generally interpreted as worsening of a disease condition.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 12
Arm/Group | Gemcabene
Number analyzed (Participants) | 0

25. Secondary Outcome: Change in Procollagen III
Description: Procollagen III peptide levels can be used to assess the degree of collagen turnover and liver fibrosis. Increases in serum concentrations of procollagen III indicate a worsening disease state.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 12
Arm/Group | Gemcabene
Number analyzed (Participants) | 0

26. Secondary Outcome: Change in Particle Size of VLDL
Description: Lipoprotein particle size will be assessed by Nuclear Magnetic Resonance (NMR). VLDL size ranges from 30-90 nanometers (nm) and is impacted by eating a meal high in fat. A linear relationship has been seen between VLDL particle size and NAFLD degree of severity.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 12
Arm/Group | Gemcabene
Number analyzed (Participants) | 0

27. Secondary Outcome: Change in Particle Size of HDL
Description: Lipoprotein particle size will be assessed by Nuclear Magnetic Resonance (NMR). HDL size ranges from 7-13 nanometers (nm). Different sizes of HDL perform different functions in the body and this study will examine how HDL particle size is altered over time by the study treatment.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 12
Arm/Group | Gemcabene
Number analyzed (Participants) | 0

28. Secondary Outcome: Change in Particle Size of LDL
Description: Lipoprotein particle size will be assessed by Nuclear Magnetic Resonance (NMR). LDL size ranges from 21-27 nanometers (nm) and is impacted by metabolic factors. This study will examine how LDL particle size is altered over time by the study treatment.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 12
Arm/Group | Gemcabene
Number analyzed (Participants) | 0

29. Secondary Outcome: Change in Particle Size of Chylomicrons
Description: The size of chylomicrons in blood will be assessed throughout the study period. Chylomicrons are lipoprotein particles comprised of primarily of triglycerides and also contain phospholipids, and proteins. The size of chylomicrons varies and typically range from 75 to 600 nanometers (nm) in diameter. Chylomicrons are larger immediately following a meal.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 12
Arm/Group | Gemcabene
Number analyzed (Participants) | 0

30. Secondary Outcome: Change in Rate of de Novo Lipogenesis (DNL)
Description: Rate of de novo lipogenesis (DNL) will be measured using stable isotope tracers. DNL is a biochemical process occurring in the liver where fatty acids are synthesized into carbohydrates. This study will examine how the rate of DNL is altered over time by the study treatment.
Time Frame: Baseline, Week 6, Week 12
Population: as for outcome 12
Arm/Group | Gemcabene
Number analyzed (Participants) | 0

31. Secondary Outcome: Absolute Change in Abdominal Visceral Fat
Description: Abdominal visceral fat was measured with the AMRA Medical body composition profile calculated from MRI images.
Time Frame: Baseline, Week 12
Population: This analysis includes participants completing 12 weeks of gemcabene.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
Liters | 0.66 (0.58)

32. Secondary Outcome: Absolute Change in Abdominal Subcutaneous Fat
Description: Abdominal subcutaneous fat was measured with the AMRA Body composition profile calculated from MRI images.
Time Frame: Baseline, Week 12
Population: This analysis includes participants completing 12 weeks of gemcabene.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
Liters | 1.30 (0.35)

33. Secondary Outcome: Change in Liver Inflammation and Fibrosis (LIF) Score
Description: LiverMultiScan by Perspectum Diagnostics is an imaging software tool that works with MRI providing a non-invasive way to diagnose liver disease. A LIF score of <1 represents a normal liver, 1-1.99 represents mild liver disease, 2-2.99 represents moderate liver disease, and a score ⩾3 represents severe liver disease.
Time Frame: Baseline, Week 12
Population: This analysis was not performed due to early termination of the study. As the milestones for study completion were not met, funding for this analysis was not available.
Arm/Group | Gemcabene
Number analyzed (Participants) | 0

34. Secondary Outcome: Absolute Change in Height
Description: Height in centimeters was measured at each study visit.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
centimeters (cm) | 0.62 (0.92)

35. Secondary Outcome: Absolute Change in Weight
Description: Weight in kilograms was measured at each study visit.
Time Frame: Baseline, Week 12
Population: This analysis includes participants completing 12 weeks of gemcabene.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
kilograms (kg) | 5.00 (1.32)

36. Secondary Outcome: Absolute Change in Body Mass Index (BMI)
Description: Body mass index (BMI) was calculated as weight (in kilograms) divided by height (in meters) squared (kg/m^2). The change in BMI between Baseline and Week 12 is presented here.
Time Frame: Baseline, Week 12
Population: This analysis includes participants completing 12 weeks of gemcabene.
Measure: Mean (Standard Deviation); unit: kilograms per meters^2 (kg/m^2)
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
kilograms per meters^2 (kg/m^2) | 1.78 (0.36)

37. Secondary Outcome: Absolute Change in Waist Circumference
Description: Waist circumference was measured in centimeters at each study visit. The change is waist circumference between Baseline and Week 12 is presented here.
Time Frame: Baseline, Week 12
Population: This analysis includes participants completing 12 weeks of gemcabene.
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
centimeters (cm) | 5.73 (6.33)

38. Secondary Outcome: Pill Count
Description: Adherence was assessed by pill counts of returned bottles. A total of 120 pills were dispensed for the 12 week study period. Taking one pill per day for 12 weeks means that 36 pills would be returned if the participant had perfect adherence. Pill counts greater than 36 mean that doses were skipped.
Time Frame: Week 12
Population: This analysis includes participants completing 12 weeks of gemcabene.
Measure: Mean (Standard Deviation); unit: Number of pills returned
Arm/Group | Gemcabene
Number analyzed (Participants) | 3
Number of pills returned | 52.0 (19.1)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and documented from the time of first dose of study drug (Study Day 1) until the Week 16 Follow-up Visit.
Arm/Group | Gemcabene
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcabene (N=6)
Increase in liver fat percentage (Hepatobiliary disorders) | 3
Increase in Creatine Kinase (General disorders) | 1
Elevated liver enzymes (Hepatobiliary disorders) | 1
Nausea (General disorders) | 1
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 1
Anxiety (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Vomitting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT03436420/Prot_SAP_000.pdf